CLINICAL TRIAL: NCT01532141
Title: Effect of Rasagiline on BIA 9-1067 Pharmacokinetics in Healthy Subjects
Brief Title: Effect of Rasagiline on BIA 9-1067 Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIA-91067-113
Record Dates: First submitted 2012-01-23; First posted 2012-02-14 (Estimated); Results first posted 2015-08-20 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-07

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; BIA 9-1067
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone; rasagiline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): Period 1: 50 mg BIA 9-1067 alone Period 2: 50 mg BIA 9-1067 1 h before a single dose of rasagiline 1 mg Period 3: 50 mg BIA 9-1067 alone concomitantly single dose of rasagiline 1 mg
  Interventions: Drug: BIA 9-1067; Drug: Rasagiline
- Group 2 (Experimental): Period 1: 50 mg BIA 9-1067 1 h before a single dose of rasagiline 1 mg Period 2: 50 mg BIA 9-1067 alone Period 3: 50 mg BIA 9-1067 alone concomitantly single dose of rasagiline 1 mg
  Interventions: Drug: BIA 9-1067; Drug: Rasagiline
- Group 3 (Experimental): Period 1: 50 mg BIA 9-1067 alone concomitantly single dose of rasagiline 1 mg Period 2: 50 mg BIA 9-1067 1 h before a single dose of rasagiline 1 mg Period 3: 50 mg BIA 9-1067 alone
  Interventions: Drug: BIA 9-1067; Drug: Rasagiline

INTERVENTIONS:
Drug: BIA 9-1067 — 50 mg BIA 9-1067 (single-dose)
  Other Names: OPC, Opicapone
Drug: Rasagiline — 1 mg rasagiline (single-dose)
  Other Names: Azilect®

SUMMARY:
The purpose of this study is to investigate the effect of rasagiline on BIA 9-1067 pharmacokinetics in healthy subjects.

DETAILED DESCRIPTION:
Single-centre, open-label, randomised, three-way crossover study consisting of 3 single-dose periods separated by a washout of 14 days or more

ELIGIBILITY:
Inclusion Criteria:

* Subjects who were able and willing to give written informed consent.
* Male or female subjects aged between 18 and 45 years, inclusive.
* Subjects of body mass index (BMI) between 18.0 and 30.0 kg/m2, inclusive.
* Subjects who were healthy as determined by pre-study medical history, physical examination, vital signs, complete neurological examination and 12-lead ECG.
* Subjects who had negative tests for HBsAg, anti-HCVAb and HIV-1 and HIV-2 Ab at screening
* Subjects who had clinical laboratory test results clinically acceptable at screening and admission to each treatment period.
* Subjects who had a negative screen for alcohol and drugs of abuse at screening and admission to each treatment period.
* Subjects who were non-smokers or ex-smokers for at least 3 months.
* (If female) She was not of childbearing potential by reason of surgery or, if of childbearing potential, she used one of the following methods of contraception: double barrier or intrauterine device.
* (If female) She had a negative pregnancy test (β-HCG) at screening and admission to each treatment period

Exclusion Criteria:

* Subjects who had a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders.
* Subjects who had a clinically relevant surgical history.
* Subjects who had any significant abnormality in the coagulation tests.
* Subjects who had any significant abnormality in the liver function tests (a case-by-case decision for any abnormality was to be discussed with the Sponsor before inclusion).
* Subjects who had a history of relevant atopy or drug hypersensitivity.
* Subjects who had a history of alcoholism or drug abuse.
* Subjects who consumed more than 14 units of alcohol a week.
* Subjects who had a significant infection or known inflammatory process at screening or admission to each treatment period.
* Subjects who had acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhoea, heartburn) at the time of screening or admission to each treatment period.
* Subjects who had received fluoxetine within 5 weeks of admission to the first period.
* Subjects who had used any other medicines within 2 weeks of admission to first period that could affected the safety or other study assessments, in the investigator's opinion.
* Subjects who had previously received BIA 9-1067.
* Subjects who have used any investigational drug or participated in any clinical trial within 90 days prior to screening.
* Subjects who have donated or received any blood or blood products within the 3 months prior to screening.
* Subjects who were vegetarians, vegans or have medical dietary restrictions.
* Subjects who could not communicated reliably with the investigator.
* Subjects who were unlikely to co-operate with the requirements of the study.
* Subjects who were unwilling or unable to give written informed consent.
* (If female) She was pregnant or breast-feeding.
* (If female) She was of childbearing potential and she did not use an approved effective contraceptive method (double-barrier, intra-uterine device) or she uses oral contraceptives.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2009-11; Primary Completion 2010-02 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Béatrice Astruc, MD, Principal Investigator — Biotrial - Human Pharmacology Unit
Locations (1):
- BIOTRIAL, Rennes, France

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3
Started | 9 | 8 | 8
Period 1 | 9 | 8 | 8
Period 2 | 8 | 8 | 8
Period 3 | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 9 | 8 | 8 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 8 | 25
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 4 | 12
  Male | 5 | 4 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Plasma Drug Concentration
Time Frame: pre-dose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 h post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- BIA 9-1067 Alone: BIA 9-1067 alone.
- BIA 9-1067 1h Before Rasagiline: BIA 9-1067 1h before Rasagiline.
- BIA 9-1067 Concomitant Rasagiline: BIA 9-1067 concomitant rasagiline.
Arm/Group | BIA 9-1067 Alone | BIA 9-1067 1h Before Rasagiline | BIA 9-1067 Concomitant Rasagiline
Number analyzed (Participants) | 25 | 24 | 24
ng/mL
  BIA 9-1067 | 647 (261) | 703 (207) | 640 (224)
  Rasagiline | NA (NA) — Rasagiline was not administered | 4.260 (1.810) | 4.299 (1.638)

2. Secondary Outcome: Time of Occurrence of Cmax (Tmax)
Description: 6-mL blood samples for the determination of plasma concentrations of BIA 9-1067 and/or rasagiline will be drawn by direct venipuncture or via an intravenous catheter into potassium ethylenediaminetetraacetic acid(EDTA)Vacutainers
Time Frame: pre-dose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 h post-dose
Measure: Median (Full Range); unit: hours
Arm/Group | BIA 9-1067 Alone | BIA 9-1067 1h Before Rasagiline | BIA 9-1067 Concomitant Rasagiline
Number analyzed (Participants) | 25 | 24 | 24
hours
  BIA 9-1067 | 3.00 [0.75 to 6.0] | 3.00 [1.0 to 6.0] | 2.50 [0.5 to 6.0]
  Rasagiline | NA [NA to NA] — Rasagiline was not administered | 0.5 [0.3 to 1.5] | 0.5 [0.3 to 1.5]

3. Secondary Outcome: AUC0-t - Area Under the Plasma Concentration-time Curve From Time 0 to Last Observed Concentration
Time Frame: pre-dose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 h post-dose
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | BIA 9-1067 Alone | BIA 9-1067 1h Before Rasagiline | BIA 9-1067 Concomitant Rasagiline
Number analyzed (Participants) | 25 | 24 | 24
ng.h/mL
  BIA 9-1067 | 1966 (831.6) | 2182 (794.2) | 2064 (827.7)
  Rasagiline | NA (NA) — Rasagiline was not administered | 3277 (1114) | 3370 (1115)

ADVERSE EVENTS:
Groups:
- Before Treatment: Before treatment.
Arm/Group | Before Treatment | BIA 9-1067 Alone | BIA 9-1067 1h Before Rasagiline | BIA 9-1067 Concomitant Rasagiline
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 3/25 | 11/25 | 4/24 | 3/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Before Treatment (N=25) | BIA 9-1067 Alone (N=25) | BIA 9-1067 1h Before Rasagiline (N=24) | BIA 9-1067 Concomitant Rasagiline (N=24)
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 2 | 1
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 6 | 1 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other